CLINICAL TRIAL: NCT05002712
Title: Effectiveness of Concurrent Training on the Performance of Team Sports Athletes
Brief Title: Concurrent Training on the Performance of Team Sports Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REC/0783 Saima Tariq
Record Dates: First submitted 2021-08-05; First posted 2021-08-12 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Sports Physical Therapy
Keywords: Concurrent training,; High resistance training,; Contrast strength training,; Elastic resistance training,; Physical performance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Heavy resistance training (Experimental): Group A
  Interventions: Other: Heavy resistance training
- Contrast strength training (Experimental): Group B
  Interventions: Other: Contrast strength training
- Elastic resistance training (Active Comparator): Group C
  Interventions: Other: Elastic resistance training

INTERVENTIONS:
Other: Heavy resistance training — Their training program included 4 resistance exercises with heavy weight lifting of the leg muscles. 3 sets of 6-8 repetitions of 80-90 % of maximal load were performed with a barbell squat (range of 0 to 90º knee flexion), lying leg curl, seated calf raises, and leg extension. The rests between the sets and the exercises lasted 5 minutes.
  Arms: Heavy resistance training
Other: Contrast strength training — Their resistance training program contained the same exercises as the high resistance training group, but with different intensity. Athlete performed each exercise for the first time with 5-7 reps with 80 % of the 1RM load followed by 15-20 reps with 40 % of the maximal load to complete the 3 sets for each exercise. The rest period between series was 60 seconds and the rest period between exercises was 5 minutes. For example, 5 heavy barbell squats followed immediately by 20 squat with lighter weight to complete 3 sets.
  Arms: Contrast strength training
Other: Elastic resistance training — During the intervention, the group conducted a 'elastic resistance training' with the same muscle groups. External resistance was provided by blue thera-band latex-free exercise bands in this training. Each exercise was performed three times for a total of 15-25 repetitions. In between sets, a 5-minute rest period was given and there was a 25-second rest period in between exercise performance. The intensity of each exercise was increased with the black thera band at the midpoint (start of week 7) of the training. The following figure shows the resistance of the blue and black bands to 100 percent elongation. Following figure shows the resistance offered by blue and black band at 100% elongation.
  Arms: Elastic resistance training

SUMMARY:
This study will add to the existing pool of knowledge with more appropriate sample size. The main purpose will be to provide coaches with a practical proposal for concurrent training(CT) to improve athletes' performance in mixed type sports and team sports. This study, therefore, will test the aspects of CT by evaluating and comparing the training adaptations induced by three forms of strength training modes in CT. One mode will be of Heavy-Resistance training where athlete will perform exercise with 80-90% of their 1RM. Second mode will be of Contrast-Strength training that will alternate the use of heavy and light resistance exercises and third mode will be Elastic Resistance Training. In the present study, these three strength protocols will be balanced for sequence of exercise, volume, duration, and other variables, so that the protocols differed only in the intensity of strength training. Comparing their training adaptations therefore will enable evaluation of the role of different forms of strength training in CT outcomes on performance.

DETAILED DESCRIPTION:
Sports performance is influenced by the interaction of several physical variables. For this reason, most sports need both strength and endurance capacities to maximize overall performance. Therefore, a combination of resistance and aerobic training, usually called concurrent training (CT), has been used recently as a way of simultaneously improving strength and aerobic performances according to the needs of a specific sport. This combination can be challenging and can influence training adaptations, being a problematic issue for coaches. Several investigators report that combined or concurrent training (CT), in which strength and aerobic endurance training are included in the same training sessions or program, interferes with the development of muscle strength or power. Reduction in strength adaptations from CT could result from neuromuscular fatigue induced by concurrent aerobic endurance exercise, which could limit the maximal muscle force that can be produced during resistance training. A converse reduction in aerobic capacity from concurrent training has seldom been reported. The reduction in strength adaptations from concurrent strength and aerobic endurance training has been termed the interference effect or phenomenon.

In contrast to interference, several investigators report compatibility of strength and endurance training, i.e., no reduction in strength adaptations from concurrent strength and aerobic endurance training. In sports applications, concurrent training has been reported to increase diverse measures of performance in basketball players, competitive rowers, endurance runners, soccer players, professional handball players, and competitive cyclists. These findings suggest that in athletes, at least, concurrent strength and aerobic endurance training has complimentary or synergic effects, rather than the contradictory or antagonistic effects implied by interference.

Therefore, clarifying the concurrent training effects is necessary and will have implications for medicine, science, sports, and recreational exercise. In sports, effects of CT i.e. interference or synergy are crucial to exercise physiologists, coaches, trainers, and athletes, who invest substantial time and resources to maximize training adaptations and competitive efficiency. Confirmation of synergy effect of CT, in contrast, could lead to more efficient athletic training protocols.

Although, some researches have de-emphasized aerobics in resistance training programs, for example, bodybuilders have portrayed aerobics as counterproductive to resistance training adaptations. On the contrary, however, several United States national certifying, training, and medical organizations recommend CT to maximize the benefits of exercise at all levels, including the American College of Sports Medicine (ACSM), the American Diabetes Association (ADA), and the National Strength and Conditioning Association (NSCA).

ELIGIBILITY:
Inclusion Criteria:

* Male athletes.
* Athletes participating in team sports.
* Those who have been new to the training and the duration of training period are not more than 03 months.

Exclusion Criteria:

* Experiencing symptoms from musculoskeletal injuries to the lower extremity.
* Any systemic pathology.
* Recent surgery.
* Participating in any other high strength/power training program during last 4 weeks of this time period.

Ages: 14 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 48 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Vertical height jump test | 6th week
  The vertical jump test measures the power of lower-body. The athlete stands horizontally against a wall and reaches out with the hand nearest to the wall for the test. The point of the extended arm's fingertips is marked when holding the feet flat on the ground. This is the height at which you can hit while standing. The athlete then takes a step away from the wall and jumps as far as possible upwards, using both arms and legs to help move the body upwards. The attempt to touch the wall at the top of the jump is recorded again. The score is the difference in distance between the two reaching heights. The best of three attempts is recorded. It is also a valid (r=0.95) and reliable tool (r=0.97). Measure the height of your highest jump and then subtract your height from highest jump in cm/inch.
1 Repetition Maximum (1RM) | 6th week
  Athletes are first advised to warm up with a light resistance that allows for 5-10 repetitions with ease. After a 1-minute rest time, a new load is determined by adding 10-20% to the warm-up load, which should allow for 3-5 repetitions. Estimate a near-maximum load that would allow for 2-3 repetitions after a 2-minute rest time by adding 10-20 percent again.
505 Agility test | 6th week
  The 505 Agility test assess your ability to turn 180 degrees. As seen in the diagram, markers are positioned 5 and 15 metres apart from a line drawn on the ground. The runner runs from the 15 metre marker to the line, through the 5 metre markers, turns on the line, and runs back through the 5 metre markers (the run in distance is to build up speed). The time is taken from when the athletes run through the 5 metre marker for the first time, and it is halted when they return through these markers (that is, the time taken to cover the 5 m up and back distance - 10 m total).
Speed of Change of Direction (COD) | 6th week
  An athlete's change of direction can also be measured by dividing his 505 time scored by 10m, the straight line distance. Formula will be: Speed of COD (m/sec) = 10m/score of 505 test in sec
30 Meter Sprint Test | 6th week
  It includes running a single maximal sprint over a distance of 30 meters, taking two time trials and recording the best time to the nearest two decimal places. Start from a stationary position, one foot in front of the other. The front foot must be either on or behind the starting line. This starting position should also be retained for 2 seconds before starting and the stopwatch should be kept ready.
YMCA Sit and Reach Test | 6th week
  The sit and reach test is a common method to evaluate lower back and hamstring flexibility. The athlete takes off his trainers, stretches and warms up properly, and then sits with his knees straight, bisecting a yardstick. The yardstick or tap is put on the floor between the subject's knees, and the heels must not move through the 15-inch section marked as 0. The athlete's hands are straight out in front of him on top of each other, and he slowly reaches out, reaching the yardstick and holding it for two seconds. The average of two trials is noted.
Yo-Yo Intermittent Recovery Test | 6th week
  The Yo-Yo test is a maximum aerobic endurance fitness test, involving running between markers 20 meters apart, at increasing speeds, until exhaustion. The Yo-Yo Intermittent Recovery Test comes in two versions: Level 1 begins at 10 km/hr and is used by younger people, and Level 2 starts at 13 km/hr.
VO2 max | 6th week
  It refers to the maximum amount of oxygen that can be used during exercise. It is widely used to measure aerobic endurance or cardiovascular fitness for athletes. Formula has been published to estimate VO2max (ml/min/kg) from Yo-Yo IR1 results and to obtain a fitness ranking.
  - Formula : VO2max (ml/min/kg) = distance run (m) × 0.0084 + 36.4

CONTACTS AND LOCATIONS:
Overall Officials: Danish Latif, MSPT-SPT, Principal Investigator — Riphah International University
Locations (1):
- Army Heritage Foundation (AHF), Ayub National Park, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No